CLINICAL TRIAL: NCT02555007
Title: Phase IA/IB of Metronomic Chemotherapy Based on Adaptative Bio-mathematical Model of Oral Vinorelbine in Patients With Non Small Cell Lung Cancer or Malignant Pleural Mesothelioma
Brief Title: Metronomic Chemotherapy Based on Adaptative Bio-mathematical Model of Oral Vinorelbine in Patients With NSCLC or MPM
Acronym: NVB Metro
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-53
Record Dates: First submitted 2015-09-11; First posted 2015-09-21 (Estimated); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Non Small Cell Lung Cancer (NSCLC); Malignant Pleural Mesothelioma (MPM)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Mesothelioma, Malignant | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral Vinorelbine (Experimental)
  Interventions: Drug: Vinorelbine

INTERVENTIONS:
Drug: Vinorelbine

SUMMARY:
Background: Metronomic oral Vinorelbine has efficacy in metastatic NSCLC and malignant Pleural Mesothelioma, but all the studies published thus far were based upon a variety of empirical and possibly suboptimal schedules, with inconsistent results. Mathematical modeling showed by simulation that a new metronomic protocol could lead to a better safety and efficacy profile.

Design: This phase Ia/Ib trial was designed to confirm safety (phase Ia) and evaluate efficacy (phase Ib) of a new metronomic oral vinorelbine schedule. Patient with metastatic NSCLC or malignant Pleural Mesothelioma, after failure of standard treatments, ECOG 0-2 and an adequate organ functions, will be eligible. Our mathematical PK-PD model suggested an alternative weekly D1, D2 and D4 innovative schedule (named Vinorelbine Theoretical Protocol) with a dynamic intake of 60, 30 and 60 mg, respectively. Trial recruitment is two-staged as 12 patients are planned to participate in the phase Ia, to confirm safety and consolidate the calibration of the average parameters of the model. Depending the phase Ia result, and after favorable decision of a consultative committee, the extension phase (phase Ib) will be an efficacy study and will include a number of 20 patients receiving the Optimal Vinorelbine Theoretical Protocol. The primary endpoint is the tolerance (assessed by CTC v4.0) for the phase Ia and the objective response according to RECIST 1.1 for the phase Ib.

An ancillary study on circulating angiogenesis biomarkers will be a subproject of the trial.

Discussion: this ongoing trial is the first to prospectively test a mathematical optimized schedule in metronomic chemotherapy. As such, this trial can be considered as a proof-of-concept study demonstrating the feasibility to run a computational-driven protocol to ensure an optimal efficacy/toxicity balance in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) ≥ 18 years of age.
* Patients with histologically documented, locally advanced or recurrent (stage IIIB) or metastatic (Stage IV) non-small cell lung Cancer or malignant pleural mesothelioma, for which no standard exits.
* Presence of at least one measurable lesion according to RECIST v.1.1 for NSCLC and modified RECIST 1.1 for MPM
* ECOG performance status ≤2

Exclusion Criteria:

* ECOG performance status >2
* Patients with significant or uncontrolled cardiovascular disease (eg, congestive heart failure, angor, arrhythmia) within 6 months of starting study treatment
* Any neurological or psychiatric condition interfering with the understanding of study
* Infectious condition uncontrolled
* Any other medical condition that would jeopardize the subject participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08-26 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Phase IA : Treatment-related hematological toxicities (neutropenia) of grade 3-4 as assessed by CTCAE v4.0 | Participants will be followed for the a maximum period of 24 months.
Phase IB : Objective response rate according to RECIST1.1 for NSCLC and RECIST1.1 modified for MPM | Participants will be followed for the a maximum period of 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Director, Study Director — Assistance Publique des Hôpitaux de Marseille
Locations (1):
- Assistance Publique des Hôpitaux de Marseille (CEPCM), Marseille, France

REFERENCES:
- [Derived] Barlesi F, Imbs DC, Tomasini P, Greillier L, Galloux M, Testot-Ferry A, Garcia M, Elharrar X, Pelletier A, Andre N, Mascaux C, Lacarelle B, Cheikh RE, Serre R, Ciccolini J, Barbolosi D. Mathematical modeling for Phase I cancer trials: A study of metronomic vinorelbine for advanced non-small cell lung cancer (NSCLC) and mesothelioma patients. Oncotarget. 2017 Jul 18;8(29):47161-47166. doi: 10.18632/oncotarget.17562. PMID 28525370